CLINICAL TRIAL: NCT02926716
Title: Efficacy of Narrow Band Imaging Technique for Identifying Resection Margin Status After Gastrectomy for Gastric Cancer
Brief Title: NBI for Identifying Resection Margin Status in Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Sang-Uk Han, Professor, Department of Surgery, Ajou University School of Medicine, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-SMP-15-10
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Gastric Cancer
Keywords: Stomach neoplasm; Endoscopy; Narrow band imaging
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
As the proportion of early gastric cancer has been steadily increased in Korea, so has function-preserving surgery. The function preserving surgery is characterized by the minimized extent of gastrectomy, so this implies that bilateral margins are getting shorter than those of standard gastrectomies.

Currently, there is only one way to identify resection margin status in gastric cancer, 'frozen biopsy'. However, it is labor-intensive and time-consuming procedure. In addition, the results rely on the pathologist's expertise, thereby it showed limitation of its accuracy; high false negative rate of signet ring cell carcinoma was reported in a previous study.

Recently, many studies on magnifying endoscopy with narrow band imaging(NBI) demonstrated that this emerging technique is useful to identify the gastric tumor margin more clearly in vivo, compared with conventional indigocarmine chromoendoscopy. So it was hypothesized that NBI may allow reliable delineation of tumor and identification of resection margin status in the specimen after gastrectomy for gastric cancer.

DETAILED DESCRIPTION:
1. Tumor delineation and identification of resection margin:

   After specimen delivery from the abdomen, frozen biopsy is performed before checking tumor margin. After inspection with NBI, the tumor margin is marked with electrocauterization. The tumor size and the lengths of both resection margins are evaluated using a ruler.
2. Pathologic examination:

The specimen is sliced as 4mm interval paralleled to the markings. Tumor size, the status of both resection margins, and microvessel density are evaluated under the 200 magnified view.

ELIGIBILITY:
Inclusion Criteria:

* The patient from over 20 to under 90 years
* The patient who is diagnosed as gastric cancer clinically by endoscopy or computed tomography
* The patient who is informed and consent about the purpose and contents of this study prior to the participation in this study

Exclusion Criteria:

* The patient who shows far advanced gastric cancer preoperatively or intraoperatively
* The patient with previous medical history of other treatment for gastric caner such as endoscopic resection, chemotherapy, radiation, immunotherapy, and so on

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient who is diagnosed as early staged gastric cancer preoperatively
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Accuracy for identifying the status of resection margin | 2 weeks
  The status of resection margin assessed by NBI during the operation is confirmed by the pathologic examination at postoperative 2 weeks

SECONDARY OUTCOMES:
Tumor size | 2 weeks
  The tumor size assessed by NBI during the operation is confirmed by the pathologic examination at postoperative 2 weeks
Microvessel density | 4 weeks
  The status of resection margin assessed by NBI during the operation is confirmed by the pathologic examination at postoperative 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University School of Medicine, Suwan, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Spicer J, Benay C, Lee L, Rousseau M, Andalib A, Kushner Y, Marcus V, Ferri L. Diagnostic accuracy and utility of intraoperative microscopic margin analysis of gastric and esophageal adenocarcinoma. Ann Surg Oncol. 2014 Aug;21(8):2580-6. doi: 10.1245/s10434-014-3669-7. Epub 2014 May 8. PMID 24806114
- [Background] Kiyotoki S, Nishikawa J, Satake M, Fukagawa Y, Shirai Y, Hamabe K, Saito M, Okamoto T, Sakaida I. Usefulness of magnifying endoscopy with narrow-band imaging for determining gastric tumor margin. J Gastroenterol Hepatol. 2010 Oct;25(10):1636-41. doi: 10.1111/j.1440-1746.2010.06379.x. PMID 20880172
- [Background] Yamada S, Doyama H, Yao K, Uedo N, Ezoe Y, Oda I, Kaneko K, Kawahara Y, Yokoi C, Sugiura Y, Ishikawa H, Takeuchi Y, Saito Y, Muto M. An efficient diagnostic strategy for small, depressed early gastric cancer with magnifying narrow-band imaging: a post-hoc analysis of a prospective randomized controlled trial. Gastrointest Endosc. 2014 Jan;79(1):55-63. doi: 10.1016/j.gie.2013.07.008. Epub 2013 Aug 7. PMID 23932092
- [Background] Eleftheriadis N, Inoue H, Ikeda H, Maselli R, Onimaru M, Yoshida A, Ito H, Hamatani S, Kudo SE. Improved optical identification of laterally spreading type "0-IIb" gastric lesion with narrow band imaging magnification endoscopy. Ann Gastroenterol. 2014;27(3):267-269. PMID 24975679
- See also: Institutional Review Board, Ajou University Hospital — https://eirb.ajoumc.or.kr